CLINICAL TRIAL: NCT01386346
Title: Phase I Study of Epigenetic Priming Using Azacitidine With Neoadjuvant Chemotherapy in Patients With Resectable Esophageal Cancer
Brief Title: Epigenetic Priming Using Azacitidine With Neoadjuvant Chemotherapy for Resectable Esophageal Cancer
Acronym: VEOX
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1012011450; VZ-ESOPH-PI-273 (Other: Celgene Corporation)
Record Dates: First submitted 2011-05-10; First posted 2011-07-01 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Esophageal Cancer; Malignant Neoplasm of Cardio-esophageal Junction of Stomach
Keywords: gastroesophageal junction; GEJ; esophageal; esophagus
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Azacitidine; Oxaliplatin; Epirubicin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects (Experimental): Azacitidine Dose level -1: 50 mg/m2 subcutaneous injection on Day 1-3 of a 21 day cycle. Repeat for a total of 3 cycles. Dose level 1: 75 mg/m2 subcutaneous injection on Day 1-3 of a 21 day cycle. Repeat for a total of 3 cycles. Dose level 2: 75 mg/m2 subcutaneous injection on Day 1-5 of a 21 day cycle. Repeat for a total of 3 cycles.
  Oxaliplatin on Day 1 130mg/m2 Epirubicin on Day 1 50mg/m2 Capecitabine 625 mg/m2
  Interventions: Drug: Azacitidine; Drug: Oxaliplatin; Drug: Epirubicin; Drug: Capecitabine

INTERVENTIONS:
Drug: Azacitidine — Dose level -1: 50 mg/m2 subcutaneous injection on Day 1-3 of a 21 day cycle. Repeat for a total of 3 cycles. Dose level 1: 75 mg/m2 subcutaneous injection on Day 1-3 of a 21 day cycle. Repeat for a total of 3 cycles. Dose level 2: 75 mg/m2 subcutaneous injection on Day 1-5 of a 21 day cycle. Repeat for a total of 3 cycles.
  Other Names: Vidaza®; 5-Azacitidine
Drug: Oxaliplatin — 130 mg/m2 IV on Day 3 or 5 of each 21 day cycle. Repeat for a total of 3 cycles.
  Other Names: Eloxatin
Drug: Epirubicin — 50 mg/m2 IV on Day 3 or 5 of each 21 day cycle. Repeat for a total of 3 cycles.
  Other Names: Ellence
Drug: Capecitabine — 625 mg/m2 orally twice daily beginning on Day 3 or 5 and will be taken without interruption for each 21-day cycle.
  Other Names: Xeolda

SUMMARY:
The purpose of this study is to see whether giving azacitidine before each cycle of chemotherapy prior to surgery is safe.

DETAILED DESCRIPTION:
Currently patients with resectable (can be removed by surgery) esophageal cancer will receive chemotherapy before surgery to try to shrink the tumor before it is removed. This study will evaluate whether giving azacitidine before each cycle of chemotherapy to increase the shrinkage of the tumor prior to surgery is safe.

Azacitidine is currently approved by the Food and Drug Administration (FDA) for treatment of myelodysplastic syndrome (MDS). Azacitidine is not approved by the FDA for use in this study and is therefore considered investigational. Because azacitidine has not been given before in combination with epirubicin, oxaliplatin and capecitabine, we will also evaluate the safety and tolerability of azacitidine and find out what dose of azacitidine is safe to give with this chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma or poorly differentiated carcinoma of the intrathoracic esophagus or gastroesophageal junction (GEJ) and deemed resectable by the thoracic surgeon.
* No prior chemotherapy for esophageal or GEJ cancer.
* ECOG Performance status 0-2.
* Adequate bone marrow, kidney and liver function.
* Ability to understand and the willingness to sign a written informed consent document.
* Subjects of child-bearing potential must agree to use effective means of contraception (men and women).
* Prior malignancy is acceptable if the subject is considered to be cured. In most cases this will mean a 5-year disease-free period.

Exclusion Criteria:

* Patients with cervical esophageal cancer or esophageal cancer with squamous cell carcinoma morphology.
* Subjects receiving any other investigational agent or received prior chemotherapy for esophageal or GEJ cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to azacitidine, epirubicin, oxaliplatin, capecitabine and mannitol.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment.
* Pregnant (positive pregnancy test) or lactating women.
* Patients with active infection, serious inter-current medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of dose limiting toxicity (DLT) | First 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No